CLINICAL TRIAL: NCT06256887
Title: SONNO - Sleep Spindles Organization as an Early Neural Marker of Neuromotor Outcome: a New, Fast, Safe, Cost-effective and Infant-friendly EEG Tool to Monitor Early Sensory-motor Function in Infants at Risk of Neuromotor Disorders.
Brief Title: Sleep Spindles Organization as an Early Neural Marker of Neuromotor Outcome
Acronym: SONNO
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Viviana Marchi, MD, PhD, IRCCS Fondazione Stella Maris
Other Study IDs: GR-2021-12375367
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: EEG Sleep Spindles; Motor Outcome; Cerebral Palsy; SMA1
Keywords: Infant; Sensorimotor Development; Automatic spindle detector; Biomarker; EEG
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infants at risk of Cerebral Palsy: N= 20, Infants at risk of Unilateral Cerebral Palsy (UCP); N= 20, Infants at risk of Bilateral Cerebral Palsy (BCP).
- Infants with diagnosis of SMA1: N=20, Infants with a diagnosis of SMA type 1.
- Infants at very low neurodevelopmental risk (control group): N=20, Infants born preterm or at term in absence of perinatal neurological complications, therefore a very low neurodevelopmental risk.

SUMMARY:
The goal of this observational study is to test the effectiveness of quantitative early biomarkers in the sleep electroencephalogram (EEG), namely sleep spindles, as predictors of early sensorimotor maturation and long-term motor outcome. Spindles are discrete events, prominent over sensorimotor areas, that reflect motor learning overnight consolidation. They represent a potential marker for the investigation of altered early sensorimotor reorganization and long-term motor outcomes in the case of neuromotor pathologies. To test this hypothesis, we will validate the prognostic accuracy of a semi-automated EEG sleep-spindles analysis in two clinical populations: 1) infants with a perinatal brain lesion, at risk of Cerebral Palsy (CP), 2) infants with Spinal muscular atrophy type 1 (SMA1), a neuromuscular disease detectable at birth with variable response to early pharmacological treatment. A group of typically developing infants (at very low neurological risk) will be enrolled in the study as control group. All participants will undergo two sleep EEG recordings at 2-5 months (T1) and 12 months (T2), respectively. Short-term neuromotor outcome will be evaluated at T1 and T2, through standard and validated assessment. Long-term neuromotor development will be defined at 18 months (T3; i.e. CP vs NO CP; SMA treatment responders vs No responders). Primary clinical and motor outcomes will be used for estimating the effectiveness of spindles' features at T1 and T2 as predictors of later clinical and motor outcomes at T3. EEG sleep features will be considered both cross-sectionally, at each time point (T1, and T2), and from a longitudinal perspective. Differences in the EEG sleep-spindle features will be evaluated within- and between-groups.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0-5 months who are at high-risk of Cerebral Palsy (CP): preterm and at term infants with a documented pre- or perinatal brain lesion at the neonatal brain MRI (i.e. hypoxic-ischemic brain injury, ischemic or hemorrhagic stroke, cystic periventricular leukomalacia, periventricular hemorrhagic infarction associated with germinal matrix-intraventricular haemorrhage);
* Infant aged 0-5 months who have received the diagnosis of SMA1, according to the perinatal genetic screening, and undergo early pharmacological treatment;
* Infants aged 0-5 months at very low neurodevelopmental risk (Control group): infants born preterm or at term in absence of perinatal neurological complications.

Exclusion Criteria (apply all groups):

* Presence of drug-resistant epilepsy or active epilepsy at T1,
* Severe sensory deficits (blindness or deafness)
* Diagnosis of progressive neurological disorders, other than SMA.

Ages: 2 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Infants at risk of Cerebral Palsy
  * Infants with diagnosis of SMA type 1
  * Infants at very low neurodevelopmental risk (control group)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Clinical dichotomous outcome | 18 (+/- 3) months
  For infants with perinatal brain damage, the primary outcome will be the diagnosis of CP: CP-YES vs CP-NO. For infants with SMA, the primary outcome will be the response to treatment: responders (SMA-R) vs non-responders (SMA-NR).
Sleep EEG (T1,T2) - quantitative sleep spindles analysis | 2-5 months, 12 (+/- 1) months
  Primary predictive measure of the study

SECONDARY OUTCOMES:
General Movements Assessment (GMA; T1) | 2-5 months
  Short-term motor outcome
Peabody Developmental Motor Scale (PDMS-II; T2 and T3) | 12 (+/- 1) months, 18 (+/- 3) months
  Long-term motor outcome
Hammersmith Infant Neurological Examination (HINE; T1, T2 and T3) | 2-5 months, 12 (+/- 1) months, 18 (+/- 3) months
  Clinical short- and long-term outcome

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Marchi, MD, PhD, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (3):
- Italy (3):
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, MI
  - IRCCS Fondazione Stella Maris, Calambrone, PI
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma

REFERENCES:
- [Background] Marchi V, Rizzi R, Nevalainen P, Melani F, Lori S, Antonelli C, Vanhatalo S, Guzzetta A. Asymmetry in sleep spindles and motor outcome in infants with unilateral brain injury. Dev Med Child Neurol. 2022 Nov;64(11):1375-1382. doi: 10.1111/dmcn.15244. Epub 2022 Apr 20. PMID 35445398